CLINICAL TRIAL: NCT06673043
Title: Anifrolumab Real-world Treatment Outcomes in Polish Patients With Systemic Lupus Erythematosus (SLE). Multicenter, Non-interventional Study
Brief Title: Anifrolumab Real-world Treatment Outcomes in Systemic Lupus Erythematosus
Acronym: SLE-ARTEMIS
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00082
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Anifrolumab; systemic lupus erythematosus; SLE; observational
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SLE Patients: Open-lable arm with SLE patients who received anifrolumab treatment in the frames of NDP in Poland.
  Interventions: Drug: Anifrolumab

INTERVENTIONS:
Drug: Anifrolumab — Anifrolumab 300 mg concentrate for solution for infusion
  Other Names: Saphnelo

SUMMARY:
The Polish multicentre observational (non-interventional) study aiming to collect data on the characteristic of patients with systemic lupus erythematosus and clinical outcomes of anifrolumab administered in the scope of routine clinical practice.

DETAILED DESCRIPTION:
This is multicenter, observational, cohort study designed to collect longitudinal data on the management and clinical outcomes of patients with SLE that received anifrolumab in the scope of routine clinical practice within the frames of National Drug Program (NDP) for up to 30 months (~ 6 months baseline and ~24 months follow-up date).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (aged ≥18 years old) patients with SLE who received anifrolumab treatment in the frames of NDP in Poland.
2. Patients willing to participate in the study and signed Informed Consent Form (ICF).

Exclusion Criteria:

1. Those who participated in anifrolumab clinical trial in the past, and/or those who participated/plans to participate in clinical trial on/after the date of first anifrolumab infusion through NDP.
2. Cognitive incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult (aged ≥18 year old) patients with SLE who received anifrolumab treatment in the frames of NDP in Poland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from index date in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score | at month 12

SECONDARY OUTCOMES:
Change from index date in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score | at month 6, 18, 24;
Change from index date in Physician Global Assessment (PGA) score | at month 6, 12, 18, 24;
Proportion of patients attaining the composite endpoint of modified SLE Responder Index (mSRI) | at month 6, 12, 18, 24;
  mSRI defined as: a reduction in SLEDAI-2K ≥4 points with no worsening in PGA ≥0.3 points
Proportion of patients attaining the composite endpoint of Lupus Low Disease Activity State (LLDAS) | at month 6, 12, 18, 24
  LLDAS defined as: SLEDAI-2K ≤4, with no activity in major organ systems and no haemolytic anaemia or gastrointestinal activity; no new lupus disease activity compared with previous assessment; PGA ≤1; current prednisone(-equivalent) dose ≤7.5mg/day; well-tolerated standard maintenance dose of immunosuppressive drugs and biologics if any.
Proportion of patients achieving the composite endpoint of remission | at month 6, 12, 18,24
  Disease activity index (cSLEDAI)=0, PGA <0.5 (0-3), prednisolone 5 mg/day or less, and stable antimalarials, immunosuppressives, and biologics.
Proportion of patients receiving antimalarials, immunosuppressives, Non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroids | every 6 months
Change from index date in corticosteroids dose | at month 6, 12, 18, 24
Proportion of steroid-free patients at every 6 months | every 6 months
Proportion of patients able to reach ≤5 mg/day of prednisolone equivalent dose at month 6, 12, 18, 24 | at month 6, 12, 18, 24
Proportion of patients with 0-25%; 26-50%; 51-75%; 76-100% glucocorticoids (GCS) dose reduction | at month 6, 12, 18, 24
Anifrolumab treatment adherence | very 6 months
  Comparison of actual and expected number of infusions (%) evaluate

CONTACTS AND LOCATIONS:
Locations (11):
- Poland (11):
  - Research Site, Bydgoszcz
  - Research Site, Bytom
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Warsaw
  - Research Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://vivli.org/